CLINICAL TRIAL: NCT05178836
Title: An Open-label, Single-arm, and Multicenter Phase Ⅱ Study to Evaluate the Efficacay and Safety of F520 Combined With F007 in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma.
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of F520 Combined With F007 in Patients With RR DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F520-101
Record Dates: First submitted 2021-12-17; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: RR DLBCL; PD-1; CD20
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F520+F007 (Experimental): Treatment period：
  F007 (375 mg/m2) administered intravenously (IV) on Day 1 of each 14-day cycle for 8 cycles.
  F520 (200mg) administered intravenously (IV) on Day 2 of each 14-day cycle for cycle 1.
  F520 (200mg) administered intravenously (IV) on Day 1 of each 14-day cycle for cycle 2 to 8.
  Maintenance period：
  F007 (375 mg/m2) administered intravenously (IV) on Day 1 of each 56-day cycle for 10 cycles.
  F520 (200mg) administered intravenously (IV) on Day 1/15/29/43 of each 56-day cycle for 10 cycles.
  Interventions: Drug: F520+F007

INTERVENTIONS:
Drug: F520+F007 — Drug: F007
  F007 is an antibody to CD20 molecules. One of the mechanisms of killing tumor cells is through antibody-dependent cell-mediated cytotoxicity (ADCC).
  Drug: F520
  F520 is a recombinant, humanized programmed death receptor-1 (PD-1) monoclonal antibody that binds to PD-1 and prevents binding of PD-1 with programmed death ligands 1 (PD-L1) and 2 (PD-L2).

SUMMARY:
This is an open-label, single-arm, and multicenter phase Ⅱ study designed to evaluate the efficacy and safety of F520 (PD-1) combined with F007(rituximab biosimilar) in patients with Relapsed/Refractory diffuse large B-cell lymphoma. About 62 patients with relapsed/refractory DLBCL plan to be enrolled in about 8 study sites of the study.

Primary objective:

The purpose is to evaluate the objective response rate of F520 combined with F007 in Relapsed/Refractory diffuse large B-cell lymphoma.

Secondary objective:

The purpose is to compare the safety of F520 combined with F007 in Relapsed/Refractory diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and ≤80 years old.
2. CD20-positive relapsed/refractory DLBCL (≥ 2 prior lines of therapy )

   Recurrence: Relapse occurred more than 6 months after the end of treatment. At least one regimen contains Rituximab.

   Refractory: Relapse within 6 months after the end of treatment or fail to reach PR after 2 treatment cycles and fail to reach CR after 4 treatment cycles. At least one regimen contains Rituximab.

   Recurrence after second-line treatment sequential autologous hematopoietic stem cell transplantation.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
4. More than 3 months life expectancy.
5. Those who agree to provide archived tumor tissue samples or fresh tissue samples
6. Biopsy confirmed CD20-positive after the last treatment. Recurrence more than 1 year needs to undergo tissue biopsy to confirm the pathological diagnosis.
7. Adequate cardiac function (LVEF≥50%).
8. At least one measurable lesion:

   For intranodal lesions, the long diameter should be >1.5cm; for extranodal lesions, the long diameter should be >1.0cm.
9. Neutrophil count (NEUT) ≥1.5×109/L and platelet count (PLT) ≥75*109/L and hemoglobin ≥75g/L, total bilirubin level (TBIL) ≤1.5×upper limit of normal (ULN), aspartic acid Aminotransferase (AST), alanine aminotransferase (ALT)≤2.5×ULN, creatinine level (Cr)≤1.5×ULN. Patients with liver metastases (TBIL≤3×ULN, ALT/AST≤5×ULN).
10. Signed an informed consent form which was approved by the institutional review board of the respective medical center.

Exclusion Criteria:

1. Primary mediastinal (thymic) large B-cell lymphoma.
2. Transformed lymphoma.
3. DLBCL invaded by special parts, such as central nervous system (CNS), testis, breast, ovary, etc.
4. High-grade B-cell lymphoma with MYC, BCL2 and/or BCL6 rearrangement.
5. History of other malignancies (except for basal/squamous cell carcinoma of the skin, in-situ carcinoma of the cervix or breast, superficial bladder cancer, lung carcinoma in situ that have been cured for more than 5 years).
6. Infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HBV-DNA titer higher than 2000 IU/mL or 1000 copies) or hepatitis C virus (HCV). Treponema pallidum (TP) antibody positive.
7. Received systemic anticancer therapy include radiation, targeted therapy, or any other anticancer therapy within 3weeks or 5 half-lives before the first administration.
8. Participation in another clinical trial in the past 4 months.
9. Received allogeneic stem cell transplantation.
10. Previous treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibody or other medications that stimulates or collaboratively inhibits T cell receptors or CAR-T.
11. Usage of immunosuppressive agents, systemic or local hormone therapy within 14 days before the first administration to achieve the purpose of immunosuppression (the daily dose is equivalent to systemic corticosteroids with prednisone> 10 mg).
12. Vaccination with an attenuated live vaccine within 4 weeks before the first administration.
13. Suffered from interstitial pneumonia in the past 6 months.
14. Severe cardiovascular disease (New York Heart Association functional class III or IV, myocardial infarction or unstable arrhythmia or unstable angina in the last 6 months, severe cardiac insufficiency, rogressive multifocal leukoencephalopathy)
15. Uncontrolled hypertension (SBP≥180mmHg and/or DBP≥100mmHg).
16. Active autoimmune diseases, including but not limited to systemic lupus erythematosus, ankylosing spondylitis, etc.
17. Severe mental illness.
18. Known hypersensitivity to any of the study drugs or its ingredients.
19. Pregnant or lactating women.
20. The researcher believes that it is not suitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Objective response rate (ORR) | 16 weeks
  To evaluate the objective response rate in patients with relapsed or refractory DLBCL.

SECONDARY OUTCOMES:
1. Complete response rate (CRR) | 16 weeks
  CR was defined as the complete disappearance of all previously detectable disease signs. CRR was percentage of participants with a CR event.
2. Progression-free survival (PFS) | 2 years
  PFS was defined as the time from randomization to first occurrence of disease progression, relapse, or death from any cause.
3. Duration of remission (DOR) | 2 years
  The time from the first assessment of complete response or partial response to the first assessment of PD or death.
4. Time to progression (TTP) | 2 years
  TTP was defined as the time from start of treatment to the date of disease progression.
5. Overall survival (OS) | 2 years
  OS defined as the time from start of treatment to the date of death due to any cause.